CLINICAL TRIAL: NCT02798991
Title: A Phase I, 14 Day, Randomized, Double-Blind (Sponsor Unblinded), Placebo-Controlled, Repeat Dose, Ascending Cohort Study to Evaluate the Safety, Tolerability Pharmacokinetics, Gastrointestinal Transit Time and Pharmacodynamic Biomarkers of GSK3179106, a REarranged During Transfection (RET) Growth Factor Receptor Tyrosine Kinase Inhibitor, in Normal Healthy Volunteers
Brief Title: A Phase I, Randomized, Placebo-controlled, Double Blind, Repeat Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Gastrointestinal Transit Time and Pharmacodynamic Biomarkers of GSK3179106 in Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205181
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: REarranged during Transfection Growth Factor Receptor Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 10 mg of GSK3179106 QD-Cohort 1 (Experimental): Eligible six subjects will receive 10 mg oral dose once daily for 14 days
  Interventions: Drug: GSK3179106
- 50 mg of GSK3179106 QD-Cohort 2 (Experimental): Eligible six subjects will receive 50 mg oral dose once daily for 14 days
  Interventions: Drug: GSK3179106
- 200 mg of GSK3179106 QD-Cohort 3 (Experimental): Eligible six subjects will receive 200 mg oral dose once daily for 14 days
  Interventions: Drug: GSK3179106
- 400 mg of GSK3179106 QD-Cohort 4 (Experimental): Eligible six subjects will receive 400 mg oral dose once daily for 14 days
  Interventions: Drug: GSK3179106
- 25 mg of GSK3179106 BID-Cohort 5 (Experimental): Eligible six subjects will receive 25 mg oral dose twice daily for 14 days
  Interventions: Drug: GSK3179106
- 200 mg of GSK3179106 BID-Cohort 6 (Experimental): Eligible six subjects will receive 200 mg oral dose twice daily for 14 days
  Interventions: Drug: GSK3179106
- Matching placebo QD-Cohort 1, 2, 3, 4 (Placebo Comparator): Eligible two subjects, per cohort, will receive oral dose of matched placebo once daily for 14 days
  Interventions: Drug: Matched Placebo
- Matching placebo BID-Cohort 5, 6 (Placebo Comparator): Eligible two subjects, per cohort, will receive oral dose of matched placebo twice daily for 14 days
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: GSK3179106 — It is uncoated round or oblong tablet with 3 strengths viz;. 5, 25 and 100 mg. It is White to slightly colored tablet and will be administered orally
  Arms: 10 mg of GSK3179106 QD-Cohort 1; 200 mg of GSK3179106 BID-Cohort 6; 200 mg of GSK3179106 QD-Cohort 3; 25 mg of GSK3179106 BID-Cohort 5; 400 mg of GSK3179106 QD-Cohort 4; 50 mg of GSK3179106 QD-Cohort 2
Drug: Matched Placebo — It is uncoated round or oblong placebo tablet prepared to match actives across all strengths. It is White to slightly colored tablet and will be administered orally
  Arms: Matching placebo BID-Cohort 5, 6; Matching placebo QD-Cohort 1, 2, 3, 4

SUMMARY:
The current study is designed to assess the safety, tolerability, pharmacokinetics (PK), gastrointestinal (GI) transit time and pharmacodynamic (PD) biomarkers of repeat oral doses of GSK3179106 administered for 14 days in normal healthy subjects. It is a randomized, double-blind, placebo-controlled, ascending cohort study. A total of 48 subjects will be randomized (8 subjects/cohort) with 3:1 allocation to GSK3179106 or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. History of regular bowel habits
* Male or Female of non-childbearing potential.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions

Exclusion Criteria:

* ALT and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1. ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Estimated Glomerular Filtration Rate <60 milliliter per minute per 1.73 square meter (mL/min/1.73m^2)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of Gastroesophageal reflux disease (GERD), dyspepsia, GI bleeding, GI surgery that could affect motility

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse event (AE) | Up to Day 25
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Cooper M, O'Connor-Semmes R, Reedy BA, Hacquoil K, Gorycki P, Pannullo K, Verticelli A, Shakib S. First-in-Human Studies for a Selective RET Tyrosine Kinase Inhibitor, GSK3179106, to Investigate the Safety, Tolerability, and Pharmacokinetics in Healthy Volunteers. Clin Pharmacol Drug Dev. 2019 Feb;8(2):234-245. doi: 10.1002/cpdd.600. Epub 2018 Sep 13. PMID 30277655